CLINICAL TRIAL: NCT06185881
Title: Clinical Performance of Short Fiber Reinforced Resin Modified Glass Ionomer Restorations Versus Resin Modified Glass Ionomer Restorations in Cervical Carious Teeth (1y Randomized Clinical Trial)
Brief Title: Clinical Performance of Short Fiber Reinforced Resin Modified Glass Ionomer Restorations in Cervical Carious Teeth (1y Randomized Clinical Trial)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rawda Hesham Abd ElAziz, Lecturer, Conservative dentistry department, Faculty of Dentistry, Cairo University., Cairo University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD 5/2022
Record Dates: First submitted 2023-12-15; First posted 2023-12-29 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Cervical Caries
Keywords: fiber reinforced glass ionomer
MeSH Terms: conditions — Root Caries

STUDY DESIGN:
Intervention Model Description: split mouth
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and both assessors will be blind to the type of material used
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short fiber reinforced resin modified glass ionomer restorations (GC Europe) (Experimental)
  Interventions: Procedure: restoration of cervical carious teeth
- Resin modified glass ionomer restoration. (Fugi II LC, GC Europe) (Active Comparator)
  Interventions: Procedure: restoration of cervical carious teeth

INTERVENTIONS:
Procedure: restoration of cervical carious teeth — restoration of carious cervical lesions by glass ionomer

SUMMARY:
This research proposal is introduced to clinically test short fiber reinforced glass ionomer material from GC Europe due to gap of knowledge present in this area. It is characterized by higher flexural strength compared to resin modified glass ionomer (RMGIC). Additionally, the short fibers provided effective toughening of the RMGIC matrix by a fiber bridging mechanism.

ELIGIBILITY:
Inclusion Criteria:

* Patients with untreated cervical carious lesions
* Patients with normal occlusion
* Vital teeth with carious cervical lesion with asymptomatic vital pulp.
* Teeth with no or minimum mobility.
* Teeth with normal occlusion.
* Teeth with surrounding healthy gingiva and supporting-structures.

Exclusion Criteria:

* Patients who are unable to return for recall appointments
* Presence of abnormal oral, medical or mental conditions.
* Patients with severe medical diseases.
* Patients with xerostomia
* Patients with parafunctional habits.
* Teeth with signs and symptoms of irreversible pulpitis or pulp necrosis.

  * Severe periodontal problems.
  * Non carious cervical lesions.

Ages: 18 Years to 38 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-12-28 (Actual)

PRIMARY OUTCOMES:
Change in Marginal integrity score | [Time Frame: Baseline, 6 months, 12 months]
  Modified USPHS criteria with Alpha, Bravo and Charlie scores (Categorical)

SECONDARY OUTCOMES:
Change in Marginal discoloration, Color match, Gross fracture scores | [Time Frame: Baseline, 6 months, 12 months]
  Modified USPHS criteria with Alpha, Bravo and Charlie scores (Categorical)
Change in Secondary caries scores | [Time Frame: Baseline, 6 months, 12 months]
  Modified USPHS criteria with Alpha and Charlie scores (Categorical)
Change in Post operative Hypersensitivity | [Time Frame: Baseline, 7 days, 6 months]
  Modified USPHS criteria with Alpha and Charlie scores (Categorical)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No